CLINICAL TRIAL: NCT00807820
Title: Phase I Study of Targeting Dominant Intraprostatic Lesion Using Functional MR Spectroscopy and High Dose Rate Brachytherapy
Brief Title: Phase I Targeting Dominant Intraprostatic Lesion Using MR Spectroscopy and HDR Brachytherapy
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H11386-24294; Grant: PC030909 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a phase I study to evaluate the feasibility and safety of using MRI/MRS to identify the dominant intraprostatic lesion (DIL) and to selectively boost the lesion using inverse planned high dose rate (HDR) brachytherapy.

The main objective is to exploit the ability of MRI/MRS to identify cancer regions within the prostate or the dominant intraprostatic lesions (DIL). The imaging data will be combined with the treatment planning CT images to define a treatment plan that will boost the dose delivered to the DIL up to 150% of the prescribed dose. Dose to the whole prostate and the dose delivered to adjacent organs will not change. This is accomplished by using inverse treatment planning software that can focus normally occurring high dose regions within the target volume to coincide with the DIL.

After enrollment, each patient will have a MRI/MRS before starting treatment. Hormonal therapy and external beam radiotherapy will be given based on current standard of practice. During HDR brachytherapy, information about the location of tumor within the prostate will be used to design the brachytherapy treatment plan. We will try to increase dose to DIL by coincide existing high dose region on DIL using inverse planning software. Dose to prostate, and adjacent structure will remain the same as the current treatment practice. Timing and the delivery of brachytherapy will not change from our current practice. After the treatment, each patient will remain on study and follow for 12 months and treatment toxicity will be evaluated. A two-stage study design will be applied with a stopping rule for safety. Once a patient comes off study he will be routinely followed for disease outcome and any late toxicities.

DETAILED DESCRIPTION:
1.1 The goal of radiotherapy is to deliver a high dose of radiation to the target volume while minimizing the dose to the surrounding normal tissue. Using CT based three-dimensional treatment planning system and multiple field technique, the three dimensional conformal radiotherapy (CRT) has become the standard of care for external beam radiotherapy for prostate cancer. Multiple institutional studies and prospective randomized trials have been done documenting the safety and efficacy of this modality. Brachytherapy is an alternative method of delivering conformal radiotherapy for treatment of prostate cancer. The technique of HDR prostate brachytherapy has been in clinical practice since the 1980's [1-13]. Kovacs et al reported one of the earliest experiences using HDR brachytherapy boost at University of Kiel.[10, 11, 13] Patients treated were mostly T2b-T3, G3. They used a combination of split course external beam radiotherapy and two 15 Gy HDR treatments. They reported 18% positive biopsy rate 18 months post treatment. The result was updated at 10 years and 78 percent of 171 patients remained free of disease at median follow-up of 55 months. Mate et al at Swedish Medical Center reported their experience with HDR brachytherapy [9]. They used a more moderated hypofractionated schema with four treatments of 3-4 Gy fractions of HDR treatments combined with 45-50 Gy of external beam radiotherapy. They recommended routine cystoscopy at the end of the implant procedure to ensure the catheters are placed at the proper depth and to avoid injuring the urethra. Pretreatment patient characteristics were stage T1b to T3c, mean initial PSA was 12.9 and Gleason grade ranges 3 to 9. They reported 84% 5-year biochemical disease free survival. Martinez et al at the William Beaumont Hospital reported the only on-going prospective dose escalation trial using HDR brachytherapy as a boost. There have been multiple updates of their results.[5-7, 12] They have continued to dose escalate using increasingly larger fractions of HDR treatment range from 5.5-6.5 Gy x 3 to 8.25-11.5 Gy x 2 combined with 46 Gy of external beam radiotherapy. As of their most recent update, they have shown acceptable toxicity level using 9.5 Gy x 2 treatments. Patients with PSA ≥ 10, T ≥ T2b, and Gleason score ≥ 7 were selected for the trial. Despite a high frequency of poor prognostic factors, the actuarial biochemical control rate was 89% at 2 years and 63% at 5 years. The 5-year actuarial rates of local failure and distant metastasis were 16% and 14%, respectively. Borghede et al. at Goteborg University in Sweden reported their experience using 50 Gy of external beam radiotherapy combined with 2 fractions of 10 Gy HDR boost.[1, 2] They used ultrasound to target tumor nodules within the prostate and gave an additional 5 Gy boost during each HDR treatment. Patients included in the study were T1-3, and grade 1-3. They report a 4% positive biopsy rate at 18-months post treatment. This is a remarkably low positive biopsy rate considering no hormonal therapy was used in the study. The results from these clinical trials and others have shown the technique of HDR brachytherapy for prostate cancer is feasible with minimal morbidity. Other institutional trials have suggested HDR boost may be more efficacious compared to external beam radiotherapy alone or external beam radiotherapy with short term hormonal therapy. Results of these studies need to be confirmed in large multi-institutional trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a candidate for HDR prostate brachytherapy
* Patient must be able to have MR scan
* Patient must have a visible DIL on MRS
* Patient has signed the protocol consent form
* No prior pelvic or prostate radiation or chemotherapy for any reason
* Induction hormonal therapy beginning ≤ 120 days prior to study entry is acceptable only if there is a MRI/MRS done prior to starting hormonal therapy
* Prostate specific antigen prior to any (hormonal) therapy must be ≤ 20 ng/ml

One of the following combinations of factors:

* Clinical stage T2a-2b, Gleason score 2-6 and PSA ≥ 10 but ≤ 20
* Clinical stage T3a-T3b, Gleason score 2-6 and PSA ≤ 20
* Clinical stage T2a-T3b, Gleason score 7-10 and PSA ≤ 20

Exclusion Criteria:

* Patient with hip prosthesis
* Patient with pacemaker
* Patient with history of radical surgery for prostate
* Patient with claustrophobia
* Patient with metal in body not safe for MR
* Stage T4 disease
* Lymph node involvement (N1)
* Evidence of distant metastases (M1)
* Previous hormonal therapy beginning > 120 days prior to registration
* Hormonal therapy prior to MRI/MRS

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient who are candidate for prostate HDR brachytherapy will be offered this protocol
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Estimate Grade 3 or greater genitourinary and gastrointestinal toxicity | One year

SECONDARY OUTCOMES:
MRI/MRS | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pouliot, Ph.D., Principal Investigator — Univerisity of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] De Bari B, Daidone A, Alongi F. Is high dose rate brachytherapy reliable and effective treatment for prostate cancer patients? A review of the literature. Crit Rev Oncol Hematol. 2015 Jun;94(3):360-70. doi: 10.1016/j.critrevonc.2015.02.003. Epub 2015 Feb 17. PMID 25819287